CLINICAL TRIAL: NCT02767310
Title: A Pivotal, Open-label, Balanced, Randomised, Two-treatment, Two-sequence, Two-period, Two-way Crossover, Single Oral Dose Bioequivalence Study of Rosuvastatin/ Verisfield 20 mg Film-coated Tablets Versus Crestor/ AstraZeneca 20 mg Film-coated Tablets in Healthy Adults Under Fasting Conditions
Brief Title: Study to Determine the Bioequivalence of Two Products Containing Rosuvastatin (20 mg/Tablet)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Verisfield UK Ltd. Greek Branch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: ROS/2016/1278
Record Dates: First submitted 2016-05-09; First posted 2016-05-10 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: Bioequivalence; two rosuvastatin-containing products
MeSH Terms: interventions — Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test Product (Experimental): Rosuvastatin 20 mg film-coated tablets
  Interventions: Drug: Rosuvastatin 20 mg film-coated tablets
- Reference product (Active Comparator): Crestor 20 mg film-coated tablets
  Interventions: Drug: Crestor 20 mg film-coated tablets

INTERVENTIONS:
Drug: Rosuvastatin 20 mg film-coated tablets — Single oral dose of 20 mg
  Arms: Test Product
Drug: Crestor 20 mg film-coated tablets — Single oral dose of 20 mg
  Arms: Reference product

SUMMARY:
The purpose of this study is to determine the bioequivalence of Rosuvastatin/ Verisfield 20 mg film-coated tablets and Crestor™/ AstraZeneca 20 mg film-coated tablets.

DETAILED DESCRIPTION:
This study aims to compare the absorption and disposition kinetics of two products containing rosuvastatin under fasting conditions. These products are: Rosuvastatin/ Verisfield 20 mg film-coated tablets, a Test product manufactured by HELP S.A., Greece and Crestor™/ AstraZeneca 20 mg film-coated tablets, a Reference product manufactured by AstraZeneca, UK. The bioequivalence of a single 20 mg dose of both products will be assessed by comparing the pharmacokinetic parameters derived from the plasma concentration-time profiles for rosuvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to provide informed consent to participate in the study.
* Comprehension of the nature and purpose of the study and willingness to comply with the requirements of the entire procedure.
* Healthy adult, human Indian volunteers within the age range of 18 to 45 years (both inclusive).
* Body Mass Index (BMI) ≥ 18.50 kg/m2 to ≤ 30.00 kg/m2.
* Hemoglobin: ≥12.0 gm% for male and ≥11.5 gm% for female.
* Absence of disease markers of HIV I & II, HBsAg, HCVAb and P24 antigen test.
* Females of childbearing age must be practicing an acceptable form of birth control for at least six months before screening, unless they have had bilateral oophorectomy or tubal ligation or their male partner has had vasectomy.
* Females of childbearing age agree to use acceptable form of birth control during the study and until the drug is washed out from the body, i.e. at least 14 days after last dosing, unless they have had bilateral oophorectomy or tubal ligation or their male partner has had vasectomy.
* Absence of significant disease or clinically significant abnormal laboratory values during the laboratory evaluations.
* Absence of any diseases in medical history or physical examination during the screening.
* Have a normal 12-lead ECG or one with abnormality considered clinically insignificant.
* Have a normal chest X-ray (P. A. view).
* Non smokers (since last six months)
* Negative serum β-HCG at the time of screening (for females only)

Exclusion Criteria:

* History / evidence of allergy or hypersensitivity to rosuvastatin or to any of the excipients or to any other drug.
* Any major illness within the last three months or any significant ongoing chronic medical illness.
* History of or active liver or kidney disease.
* History of or active deep vein thrombosis and thromboembolic disorders.
* History of breast cancer, endometrial cancer or other estrogen-dependent neoplasia, endometriosis and undiagnosed vaginal bleeding (for females only).
* History of drug abuse (including barbiturates, benzodiazepines, opioids, cocaine, cannabinoids and amphetamine etc.) within the last three months.
* History of neuropsychiatric diseases.
* History of hypothyroidism.
* Personal or family history of hereditary muscular disorders.
* History of myopathy.
* History of myalgia.
* History of rhabdomyolysis.
* History of alcohol abuse.
* History of proteinuria.
* Asian population (except Indian).
* History of interstitial lung disease.
* History of or current gastro-intestinal diseases influencing drug absorption.
* History of alcoholism (more than two years), moderate drinkers (more than three drinks per day).
* Participation in any clinical trial within last three months.
* History of difficulty with donating blood or difficulty in accessibility of veins in left or right arm.
* Donation of blood (one unit or 350 mL or more) within last three months.
* Use of any prescription drug therapy within last two weeks and over the counter (OTC) drugs or herbal products within last one week.
* Pregnant women.
* Breast feeding women.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration (AUC0-t) from zero (0) hours to time (t) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.00, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The area under the plasma concentration versus time curve, from time zero (0) to t hours
Maximum concentration (Cmax) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Maximum measured plasma concentration

SECONDARY OUTCOMES:
Time to maximum concentration (Tmax) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Time of the maximum measured plasma concentration. If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value
Elimination rate constant (Kel) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  Apparent first-order elimination or terminal rate constant
Terminal half life (t1/2) | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The elimination or terminal half-life
Area under the plasma concentration (AUC0-infinity) from zero (0) hours to infinity | Before dosing (0 hour) and 0.25, 0.50, 0.75, 1.50, 2.00, 2.50, 3.00, 3.50, 4.00, 4.50, 5.00, 6.00, 7.00, 8.00, 10.00, 12.00, 16.00, 24.00, 36.00 and 48.00 hours post-dose
  The area under the plasma concentration versus time curve from time (0) to infinity
Number of participants with Adverse Events | 6 days

CONTACTS AND LOCATIONS:
Overall Officials: Kathiria Jayesh, M.D., Principal Investigator — Synchron Research Services Pvt. Ltd.
Locations (1):
- Synchron Research Services Pvt. Ltd., Ahmedabad, Gujarat, India